CLINICAL TRIAL: NCT00052598
Title: Phase I/II Study of Adoptive Immunotherapy With CD8+ Proteinase 3 (Myeloblastin)-Specific CTL Clones for HLA-A2+ Patients With Relapse or Progression of Disease After Allogeneic Hematopoietic Stem Cell Transplant for High Risk Myeloid Leukemias
Brief Title: Therapeutic Allogeneic Lymphocytes and Aldesleukin in Treating Patients With High-Risk or Recurrent Myeloid Leukemia After Undergoing Donor Stem Cell Transplant
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1671.00; NCI-2010-00826 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA018029 (NIH)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Blastic Phase Chronic Myelogenous Leukemia; Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Blast Crisis; Leukemia, Myeloid, Acute | interventions — aldesleukin; Interleukin-2; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (adoptive immunotherapy) (Experimental): Patients receive allogeneic CD8+ PR3-specific CTLs IV over 1-2 hours on days 0, 7, 14, 28, and 49 and aldesleukin SC twice daily on days 28-41 and 49-63 in the absence of unacceptable toxicity.
  Interventions: Biological: therapeutic allogeneic lymphocytes; Biological: aldesleukin; Other: laboratory biomarker analysis; Other: flow cytometry

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes — Given IV
  Other Names: ALLOLYMPH
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Other: laboratory biomarker analysis — Correlative studies
Other: flow cytometry — Correlative studies

SUMMARY:
This phase I/II trial is studies the side effects of giving therapeutic allogeneic lymphocytes together with aldesleukin and to see how well it works in treating patients with high-risk or recurrent myeloid leukemia after undergoing donor stem cell transplant. Biological therapies, such as therapeutic autologous lymphocytes, may stimulate the immune system in different ways and stop cancer cells from growing. Aldesleukin may stimulate the white blood cells to kill cancer cells. Giving therapeutic autologous lymphocytes together with aldesleukin may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and potential toxicities associated with infusing donor CD8+ cytotoxic T lymphocytes (CTL) clones specific for Proteinase 3 (Myeloblastin) in patients with relapse/progression of high risk myeloid leukemias after transplant.

SECONDARY OBJECTIVES:

I. To determine the in vivo persistence of transferred T cells and assess migration to the bone marrow, a predominant site of leukemic relapse.

II. To determine if adoptively transferred proteinase 3 (PR3)-specific T cells mediate antileukemic activity.

OUTLINE:

Patients receive allogeneic CD8+ PR3-specific CTLs intravenously (IV) over 1-2 hours on days 0, 7, 14, 28, and 49 and aldesleukin subcutaneously (SC) twice daily on days 28-41 and 49-63 in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up every 1-3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing allogeneic hematopoietic stem cell transplantation for chronic myelogenous leukemia (CML) in accelerated or blast phase, acute myeloid leukemia (AML) beyond first remission, primary refractory AML, therapy-related AML at any stage, or acute leukemia at any stage arising in a patient with an antecedent diagnosis of a myelodysplastic or myeloproliferative syndrome (including chronic myelomonocytic leukemia, CML, polycythemia vera, essential thrombocytosis, and agnogenic myeloid metaplasia with myelofibrosis)
* Patients and donors must both be human leukocyte antigen (HLA)-A2 positive
* Patients must be able to provide blood and bone marrow samples required for this protocol
* Eligibility for Prophylactic Treatment with CD8+ CTL After Transplant (Highest Risk Subgroup):
* At time of planned treatment, CD8+ CTL specific for PR3 must have been generated and have completed Quality Control (QC) testing
* Patients must have had > 5% morphologic blasts detectable in bone marrow or peripheral blood just prior to or at the time of transplant
* Patients must have evidence of posttransplant recovery of normal hematopoiesis (absolute neutrophil count [ANC] > 500/mm^3) for at least 7 days prior to the initiation of CTL infusions
* Patients on immunosuppressive therapy for graft-versus-host disease (GVHD) are eligible for treatment if not receiving corticosteroids or if the dose of corticosteroids can be tapered to < the equivalent of 0.5 mg/kg/day of prednisone; The patient's symptoms have to remain stable and unlikely to increase to stage III or IV acute GVHD or chronic GVHD is unlikely to progress following the change in immunosuppressive therapy, after an appropriate monitoring period, as deemed by the patients treating physician and the principal investigator
* Eligibility for Treatment with CD8+ CTL at the Time of Relapse After Transplant (All Others):
* At time of planned treatment, CD8+ CTL specific for PR3 must have been generated and have completed Quality Control (QC) testing
* Patients must have evidence of recurrent/progressive disease posttransplant
* Morphologic relapse defined as one or more of the following: abnormal peripheral blasts in absence of growth factor therapy, abnormal bone marrow blasts > 5% of nucleated cells, extramedullary chloroma or granulocytic sarcoma
* Flow cytometric relapse defined as the appearance in the peripheral blood or bone marrow of cells with an abnormal immunophenotype detected by flow cytometry that is consistent with leukemia recurrence/progression
* Cytogenetic relapse/progression defined as the appearance in one or more metaphases from bone marrow or peripheral blood cells of either a non-constitutional cytogenetic abnormality identified in at least one cytogenetic study performed prior to transplant or a new abnormality known to be associated with leukemia; (for CML), an increase in the number of Ph+ metaphases from bone marrow or peripheral blood between two consecutive samples after engraftment, or an increase in the percentage of BCR/ABL+ cells by fluorescence in situ hybridization (FISH) between two consecutive samples after engraftment
* Molecular relapse/progression defined as a polymerase chain reaction (PCR) assay of bone marrow (BM) or peripheral blood mononuclear cells (PBMC) positive for the presence of the BCR/ABL messenger ribonucleic acid (mRNA) fusion transcript that quantitatively increases by greater than one order of magnitude on a subsequent sample
* Patients on immunosuppressive therapy for GVHD at the time of relapse are eligible for treatment if not receiving corticosteroids or if the dose of corticosteroids can be tapered to < the equivalent of 0.5 mg/kg/day of prednisone; the patient's symptoms have to remain stable and unlikely to increase to stage III or IV acute GVHD or chronic GVHD is unlikely to progress following the change in immunosuppressive therapy, after an appropriate monitoring period, as deemed by the patient's treating physician and the principal investigator

Exclusion Criteria:

* Exclusions for Treatment at the Time of Relapse/Progression After Transplant:
* Patients for whom CD8+ CTL clones specific for PR3 have not been generated by the time of disease relapse/progression post-transplant; these patients can potentially be treated later if CTL become available; patients whose malignant cells do not overexpress PR3, based on direct analysis of a bone marrow sample with > 50% blasts or of leukemia cells isolated for expression analysis; in either case, patients will be informed about the availability of other treatment protocols for which they might be eligible
* Patients with Karnofsky performance status or Lansky play score =< 30%
* Patients with current stage III or IV GVHD unresponsive to therapy or requiring therapy with anti-CD3 mAb, prednisone > 0.5 mg/kg/day (or corticosteroid equivalent), or other treatments resulting in the ablation or inactivation of T cells (such as other anti-T cell monoclonal antibodies); although the concurrent use of cyclosporine, FK506, or mycophenolate mofetil (MMF) is not strictly an exclusion criterion, attempts should be made to discontinue it if possible
* Patients requiring concurrent therapy with hydroxyurea or other agents that may interfere with the function or survival of infused CTL clones
* Patients with a preexisting nonhematopoietic organ toxicity that is deemed by the principal investigator to place the patient at unacceptable risk for treatment on the protocol
* Patients with graft rejection or failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2002-09; Primary Completion 2009-11 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Toxicity rate associated with infusing donor CD8+CTL clones specific for PR3 | From the first CTL infusion to 4 weeks after the final dose of CTL or IL-2

SECONDARY OUTCOMES:
In vivo persistence of transferred T-cells and assessment of migration to the bone marrow | Baseline and days +7, +11, +14, +21, and +28 after each CTL infusion
Duration of response as assessed by PCR or cytogenetic analysis of peripheral blood and bone marrow samples | Days +0, +15, +29, +50, +63, and at approximately 1 month after completion of all therapy
Proportion of responders | Approximately one month after completion of all therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Ragnarsson, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States